CLINICAL TRIAL: NCT05271825
Title: Broadband Amplification as Tinnitus Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Mie Joergensen, PhD student, Technical University of Denmark
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 766041
Record Dates: First submitted 2022-02-16; First posted 2022-03-09 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Broadband amplification (Experimental): broadband amplification: (125 Hz to 10 kHz)
  Interventions: Device: Broadband amplification from hearing aids
- Band-limited amplification (Placebo Comparator): band-limited amplification (125 Hz to 3-4 kHz)
  Interventions: Device: Band-limited amplification from hearing aids

INTERVENTIONS:
Device: Broadband amplification from hearing aids — Amplification from 125 Hz to 10 kHz
  Arms: Broadband amplification
Device: Band-limited amplification from hearing aids — Amplification from 25 Hz to 3-4 kHz
  Arms: Band-limited amplification

SUMMARY:
* The effect of broadband amplification was tested in a double-blinded crossover study
* Its effect was compared to an active placebo treatment
* An improvement in tinnitus distress was found after use of broadband amplification
* No effect was found on the tinnitus loudness

DETAILED DESCRIPTION:
This study investigated the effect of broadband amplification (125 Hz to 10 kHz) as tinnitus treatment for participants with high-frequency hearing loss and compared these effects with an active placebo condition using band-limited amplification (125 Hz to 3-4 kHz). A double-blinded crossover study. 23 participants with a high-frequency (≥ 3 kHz) hearing loss and chronic tinnitus were included in the study and 17 completed the full treatment protocol. Two different hearing aid treatments were provided for 3 months each: broadband amplification that provided gain in the frequency range from 125 Hz to 10 kHz and band-limited amplification that only provided gain in the low frequency range (≤ 3-4 kHz). The effect of the two treatments on tinnitus distress was evaluated with the Tinnitus Handicap Inventory (THI) and the Tinnitus Functional Index (TFI) questionnaires. The effect of the treatment on tinnitus loudness was evaluated with a visual analog scale (VAS) for loudness and a psychoacoustic loudness measure. Furthermore, the tinnitus annoyance was evaluated with a VAS for annoyance. The tinnitus pitch was evaluated based on the tinnitus likeness spectrum.

ELIGIBILITY:
Inclusion Criteria:

* Chronic tinnitus
* hearing thresholds (<=25 dB HL) up to 2000 Hz and hearing loss at frequencies above 2 kHz
* inexperienced hearing aid user

Exclusion Criteria:

* objective or pulsatile tinnitus
* Ménière's disease, otosclerosis, stapedectomy, stapedotomy or tympanoplasty

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory | 3 months
  Questionnaire assessing tinnitus related distress. 25 questions that can be answered with yes(4 points), sometimes (2 points), no (0 points)
Tinnitus Functional Index | 3 months
  Questionnaire assessing tinnitus related distress. 25 questions that can be answered with likert scale from 0-10 (or 0-100%) where 10 is the most extreme negative value

SECONDARY OUTCOMES:
Tinnitus loudness | 3 months
  Psychoacoustic measurement. Participants are asked to match the loudness of their tinnitus to either a pure-tone or noisy sound. The loudness of the matched tone could be changed in 3 decibel steps.
Tinnitus spectrum | 3 months
  The tinnitus spectrum rating method was adapted from Noreña et al. (2002). As the stimuli, either 2-s long pure tones (1st condition) or 2-s long 1/3-octave noise bands (2nd condition) with center frequencies ranging from 125 Hz to 14 kHz were used. The stimuli were presented monaurally via headphones to the ear corresponding to the loudest tinnitus perception. In case the tinnitus percept was the same in both ears, the stimuli were presented to the ear with the lowest average high-frequency thresholds. All stimuli were presented at the level matched to the tinnitus loudness for a 1 kHz pure tone, but always at or above 10 dB sensation level (SL).
Visual Analog Scale - annoyance | 3 months
  Likert scale from 0-10 where 0 = "My tinnitus is not annoying" and 10 = "My tinnitus is extremely annoying"
Visual Analog Scale - loudness | 3 months
  Likert scale from 0-10 where 0 = "I cannot hear my tinnitus" and 10 = "My tinnitus is extremely loud"

CONTACTS AND LOCATIONS:
Overall Officials: Mie Jørgensen, Principal Investigator — Technical University of Denmark
Locations (1):
- Technical University of Denmark, Kongens Lyngby, Denmark

IPD SHARING:
Plan to Share IPD: No